CLINICAL TRIAL: NCT01123174
Title: Effectiveness of a "Case Management Algorithm" After a Suicide Attempt in Terms of Repetition of the Suicidal Behaviors and Medico-economic Impact
Brief Title: Effectiveness of a Case Management Algorithm: ALGOS After a Suicide Attempt
Acronym: ALGOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2009_25; PHRC 2009/1902 (Other: DHOS); 2009-A00893-54 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2010-03-18; First posted 2010-05-14 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Suicide, Attempted
Keywords: Suicide; case management algorithm; suicidal behaviors; prevention of suicide
MeSH Terms: conditions — Suicide, Attempted; Suicide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALGOS group (Experimental): Algorithm of case management over the 6 months following the suicidal gesture (systematic telephone contact, postcards and crisis card)
  Interventions: Behavioral: ALGOS algorithm of case management
- Control group (No Intervention): Treatment as usual (referral back to the general practitioner)

INTERVENTIONS:
Behavioral: ALGOS algorithm of case management — If the subject survives one 1st SA (first attempter): he leaves the center where he was included with a "chart resource" (crisis card) which contains addresses of the Web sites of associations of prevention of the suicide, as well as an accessible phone number 24/24h.
  If the subject is not a first attempter : he will be recontacted on the telephone between the 10th and the 21st day following the SA. If the subject is not contacted or little observing in the plan of care, it will receive a series of postcards then regularly, with 4 recoveries: to 2, 3, 4 and 5 months after the attempt.
  Other Names: ALGOS Group
  Arms: ALGOS group

SUMMARY:
The suicidal behaviors are phenomena eminently multifactorial. It is thus always difficult to define univocal strategies of prevention of suicide repetition, during the emergency stay, i.e. almost in general population. One find 23 clinical trials in this topic in the past 25 years, and 18 are negative. The majority of the positive trials have the concern of being dissociated from an assumption of responsibility of care strictly speaking, to adopt a position "méta", nearer to the concept of "case management": how to remain in contact with the suicide attempter, without forcing it in this every day life, replacing a possible proposing, but assumption of responsibility resources reliable and quickly accessible in the event of at risk situation? Each one of these studies tests devices which seem more appropriate to such or such characteristic of this population, by retaining only simple criteria like the sex, the number of former suicide attempts, the proposal or not for an assumption of responsibility of care, the observance or not with the plan of care. Thus, it would seem interesting to combine these approaches in an algorithm entitled "ALGOS".

Main aim: To test the effectiveness of this algorithm of case management, named "ALGOS", in reducing the number of death by suicide, in terms of reduction of suicide re-attempts and the number of loss of contact patients in the ALGOS group during 6 months period, compared to a control group of suicide attempters treated as usual (i.e. primarily transmitted to the attending physician).

Secondary objectives: To evaluate, according to the method validated by Beecham in 1992, direct medico-economic impact in the year which follows the introduction of algorithm ALGOS. Reduction of the other suicidal behaviors in 6 months (reduction in the full number of suicidal repetitions in each group, evolution of the score of suicidal ideation, etc…). To evaluate the effect of the algorithm, at the 13th month. To study the possible differences within the time in terms of suicidal repetitions in the 2 groups. To propose different profiles of answers according to psychopathology, the number of suicide attempts, suicidal character, the sex,…

Methodology: Comparative simple blind prospective multicentric controlled study

DETAILED DESCRIPTION:
Evaluations: The subjects will be included in the participating centers following a suicide attempt (SA). After checking of the criteria, information and signature of the study consent, the subjects will be randomized in one of the 2 groups (ALGOS versus Control). A fax of inclusion will be sent to the centralized research team of the Clinical Investigation Center (CIC) of Lille. All the subjects included will be then evaluated at the 6th month and 13th month after the SA, during a phone call. The final evaluation will be carried out in the current of the 13th month, so as to avoid a recontact at the time of the period birthday, too charged affectively at the majority with the patients. This phone call, personal, will be carried out by an trained psychologist. A mail preventing the subject of the call will be addressed approximately 10 days before. During the evaluations at the 6th month and 13th month, the number of suicidal repetitions will be reported, consumption of care since inclusion will be noted, the scale of suicidal ideation of Beck assessed, and a psychopathological evaluation carried out (Mini International Neuropsychiatric Interview DSM IV).

ELIGIBILITY:
Inclusion Criteria:

* Surviving to a suicide attempt (SA) directly leaving the Emergency unit or have been hospitalized less than 7 days

Exclusion Criteria:

* recidivists who made 4 SA and more in the 3 past years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1040 (Actual)
Dates: Start 2010-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Number of suicide re-attempters | six months
  the number of suicide re-attempters 6 months following the attempt index

SECONDARY OUTCOMES:
Number of deaths per suicide | six months and 13 months
  Number of suicide re-attempts in the 6 months following the attempt index
Number of lost to follow up | six months and 13 months
Number of suicide re-attempters | 13 months
Number of suicide re-attempts | six months and 13 months
  Number of suicide re-attempts in the 6 months following the attempt index
Suicidal ideation intensity | six months and 13 months
  The suicidal ideation will be measured by Scale of Suicidal Ideation (A. Beck, M. Kovacs, and A. Weissman, 1979) in the 6 months following the attempt index and in the 13 months.
medical cost | six months and one year
  Numbers of hospitalisations, numbers of consultations, and drugs consummation during the year following the suicide attempt will be measured to estimate the medical cost
Evaluation of the psychopathological profile | six months and 13 months
  The psychopathological profile will be evaluated by the French version of Mini International Neuropsychiatric Interview (DSM IV)

CONTACTS AND LOCATIONS:
Overall Officials: Guillauma VAIVA, Principal Investigator — University Hospital, Lille; Michel WALTER, Principal Investigator — University Hospital, Brest
Locations (23):
- France (23):
  - University Hospital, Angers, Angers
  - General Hospital, Boulogne sur Mer, Boulogne-sur-Mer
  - University Hospital, Brest, Brest
  - University Hospital, Caen, Caen
  - University Hospital, Clermont Ferrand, Clermont-Ferrand
  - Henri Mondor Hospital, Creteil, Créteil
  - General Hospital, Douai, Douai
  - General Hospital, Dunkerque, Dunkirk
  - Health Centre Henin Beaumont, Hénin-Beaumont
  - University Hospital, Lille, Lille
  - University Hospital, Marseille, Marseille
  - General Hospital, Montauban, Montauban
  - University Hospital, Montpellier, Montpellier
  - University Hospital, Nancy, Nancy
  - University Hospital, Nantes, Nantes
  - University Hospital, Nice, Nice
  - Georges Pompidou European Hospital, Paris, Paris
  - General Hospital, Quimper, Quimper
  - University Hospital, Rennes, Rennes
  - General Hospital, Roubaix, Roubaix
  - University Hospital, Toulouse, Toulouse
  - General Hospital, Tourcoing, Tourcoing
  - General Hospital, Vannes, Vannes

REFERENCES:
- [Background] Vaiva G, Vaiva G, Ducrocq F, Meyer P, Mathieu D, Philippe A, Libersa C, Goudemand M. Effect of telephone contact on further suicide attempts in patients discharged from an emergency department: randomised controlled study. BMJ. 2006 May 27;332(7552):1241-5. doi: 10.1136/bmj.332.7552.1241. PMID 16735333
- [Background] Carter GL, Clover K, Whyte IM, Dawson AH, D'Este C. Postcards from the EDge project: randomised controlled trial of an intervention using postcards to reduce repetition of hospital treated deliberate self poisoning. BMJ. 2005 Oct 8;331(7520):805. doi: 10.1136/bmj.38579.455266.E0. Epub 2005 Sep 23. PMID 16183654
- [Background] Evans J, Evans M, Morgan HG, Hayward A, Gunnell D. Crisis card following self-harm: 12-month follow-up of a randomised controlled trial. Br J Psychiatry. 2005 Aug;187:186-7. doi: 10.1192/bjp.187.2.186. PMID 16055834
- [Background] Vaiva G, Walter M, Al Arab AS, Courtet P, Bellivier F, Demarty AL, Duhem S, Ducrocq F, Goldstein P, Libersa C. ALGOS: the development of a randomized controlled trial testing a case management algorithm designed to reduce suicide risk among suicide attempters. BMC Psychiatry. 2011 Jan 2;11:1. doi: 10.1186/1471-244X-11-1. PMID 21194496
- [Derived] Demesmaeker A, Chazard E, Vaiva G, Amad A. Risk Factors for Reattempt and Suicide Within 6 Months After an Attempt in the French ALGOS Cohort: A Survival Tree Analysis. J Clin Psychiatry. 2021 Feb 18;82(1):20m13589. doi: 10.4088/JCP.20m13589. PMID 33999539
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Vaiva G, Berrouiguet S, Walter M, Courtet P, Ducrocq F, Jardon V, Larsen ME, Cailhol L, Godesense C, Couturier C, Mathur A, Lagree V, Pichene C, Travers D, Lemogne C, Henry JM, Jover F, Chastang F, Prudhomme O, Lestavel P, Gignac CT, Duhem S, Demarty AL, Mesmeur C, Bellivier F, Labreuche J, Duhamel A, Goldstein P. Combining Postcards, Crisis Cards, and Telephone Contact Into a Decision-Making Algorithm to Reduce Suicide Reattempt: A Randomized Clinical Trial of a Personalized Brief Contact Intervention. J Clin Psychiatry. 2018 Sep 25;79(6):17m11631. doi: 10.4088/JCP.17m11631. PMID 30256552